CLINICAL TRIAL: NCT02439294
Title: Impact of the Obstructive Sleep Apnea Syndrome (OSAS) on the Ventricular Remodeling After Acute Myocardial Infarction
Acronym: SAS-IDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9541
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Recent Acute Myocardial Infarction
Keywords: Recent acute myocardial infarction; Obstructive sleep apnée (syndrome); Ventricular remodeling; Continuous Positive Airway Pressure
MeSH Terms: conditions — Syndrome; Ventricular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Without Obstructive Sleep Apnea (syndrome) (Other): Subjects will be randomized after the results of the polysomnography (21st day ± 10) in one of this three groups
  Interventions: Other: Without Obstructive Sleep Apnea (syndrome)
- Mild or moderate Obstructive Sleep Apnea (syndrome) (Other): Subjects will be randomized after the results of the polysomnography (21st day ± 10) in one of this three groups
  Interventions: Other: Mild or moderate Obstructive Sleep Apnea (syndrome)
- Severe Obstructive Sleep Apnea (syndrome) (Other): Subjects will be randomized after the results of the polysomnography (21st day ± 10) in one of this three groups
  Interventions: Other: Severe Obstructive Sleep Apnea (syndrome); Device: CPAP

INTERVENTIONS:
Other: Without Obstructive Sleep Apnea (syndrome)
  Arms: Without Obstructive Sleep Apnea (syndrome)
Other: Mild or moderate Obstructive Sleep Apnea (syndrome)
  Arms: Mild or moderate Obstructive Sleep Apnea (syndrome)
Other: Severe Obstructive Sleep Apnea (syndrome)
  Arms: Severe Obstructive Sleep Apnea (syndrome)
Device: CPAP
  Arms: Severe Obstructive Sleep Apnea (syndrome)

SUMMARY:
Coronary artery disease is a common and serious disease, the leading cause of death worldwide. Obstructive sleep apnea syndrome (OSAS) is common and often under-diagnosed in coronary artery disease where it could be involved in the pathophysiology and perhaps prognosis. The entanglement of the two pathologies is actually quite well known, in particular the consequences of one over the other just beginning to be studied. Understanding the pathophysiology through new imaging modalities should improve the management of patients to propose new approaches.

"SAS-IDM" is an interventional and prospective study conducted at the University Hospital of Montpellier. Patients will be divided in three groups depending of the results of the polysomnography: 1/ AHI < 5/h: normal, without OSA ; 2/ 5/h ≤ AHI < 30/h: mild or moderate OSA ; 3/ IAH ≥ 30/h: severe OSA. A treatment by CPAP will be proposed to patients of the group "severe OSA".

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures,
* Adults, men and women aged < 90 years,
* Hospitalized in Intensive Care Units, MI confirmed by the study of the coronary arteries (coronary angiography) in acute phase (primary coronary angiography) or secondarily (ambulatory IDM IDM initially reperfused by thrombolysis),
* Myocardial infarction defined the criteria normally applied (STEMI: ST segment depression greater than 2 mm in at least 2 contiguous leads or new onset of pain and a left bundle branch block),
* The score of delayed enhancement MRI should be greater than 5 segments of 17 during the first MRI (criterion of severity of AMI),
* The subject must be affiliated to a social security scheme

Exclusion Criteria:

* Patients for whom CPAP equipment has demonstrated its usefulness regardless of cardiovascular context

  * Patients sleepy (Epworth score> 13)
  * Road Truckers
* Contraindication to achieve cardiac MRI (primary endpoint):

  * known and crippling claustrophobia,
  * metal clips intracranial, intraocular,
  * presence of an implantable defibrillator
  * presence of a pacemaker
  * history of injury by firearm or shrapnel balance without known projections
  * hypersensitivity to gadolinium products (or history of systemic sclerosis skin) or severe renal impairment with creatinine clearance <30 ml / min
  * any other known cause of contra-indication.
* Mild infarction (rate of late enhancement MRI in less than or equal to 4 segments of 17 during the first MRI)
* Patient previously treated with CPAP prior MI or already experienced with sleep apnea syndrome.
* SAS whose central part is predominantly (> 50%)
* General

  * Inability to understand the nature and goals of the study and / or communication difficulties with the investigator
  * No affiliation to a French social security recipient or not such a scheme
  * Major protected by law (guardianship, curators or under judicial protection)
  * deprivation of liberty by judicial or administrative decision
  * Increased likelihood of non compliance to the protocol or abandonment under study
  * History or presence of psychoactive substance abuse
  * pregnancy, become pregnant, or breastfeeding

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Changes in diameter (mm) and end diastolic and systolic LV volumes (mL) at 6 months of acute MI among a group of patients without OSA (AHI <5 / h) and a group of patients with mild to moderate OSA (AHI between 5 and 30 / h) | 6 months of acute MI
Transmural enhancement (%) at 6 months of acute MI among a group of patients without OSA (AHI <5 / h) and a group of patients with mild to moderate OSA (AHI between 5 and 30 / h) | 6 months of acute MI
Thickness of the LV wall (mm) at 6 months of acute MI among a group of patients without OSA (AHI <5 / h) and a group of patients with mild to moderate OSA (AHI between 5 and 30 / h) | 6 months of acute MI
Presence no reflow at 6 months of acute MI among a group of patients without OSA (AHI <5 / h) and a group of patients with mild to moderate OSA (AHI between 5 and 30 / h) | 6 months of acute MI

SECONDARY OUTCOMES:
The difference in cardiac remodeling in cardiac MRI at 6 months between the three diagnostic categories | At 6 months after inclusion
The difference in cardiac remodeling in cardiac MRI between the date of inclusion and 6 months between diagnostic categories. | Between the date of inclusion and 6 months
The difference of left ventricular remodeling in cardiac MRI between the date of inclusion and 6 months in the severe OSA group based on the assumption (good compliance and effectiveness of PPC or not) | Between the date of inclusion and 6 months
The occurrence of cardiovascular events during the first year following the IDM depending on the initial AHI index. | Between the date of inclusion and one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Arnaud de Villeneuve - CHU de Montpellier, Montpellier, France